CLINICAL TRIAL: NCT01402505
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES): Laparoscopic Assisted Trans-Vaginal Sleeve Gastrectomy
Brief Title: Transvaginal NOTES Sleeve Gastrectomy
Status: Withdrawn | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Other Study IDs: 081036, 141812
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: obesity; sleeve gastrectomy; transvaginal NOTES
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Transvaginal NOTES sleeve gastrectomy: Transvaginal NOTES sleeve gastrectomy
  Interventions: Procedure: Transvaginal NOTES sleeve gastrectomy

INTERVENTIONS:
Procedure: Transvaginal NOTES sleeve gastrectomy — transvaginal NOTES sleeve gastrectomy

SUMMARY:
This is a prospective chart review/data collection study of natural orifice translumenal endoscopic surgery (NOTES) for sleeve gastrectomy, that will include questionnaires administered throughout the study. Subjects enrolled will be those intending to have a transvaginal NOTES sleeve gastrectomy. Data will be collected and reviewed through 12 months post-op.

ELIGIBILITY:
Inclusion:

1. Diagnosis of morbid obesity BMI > 40
2. Female, age 18-75
3. Mentally competent to give informed consent
4. Scheduled to undergo a transvaginal NOTES sleeve gastrectomy

Exclusion:

1. Pregnant women
2. BMI < 40

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-75 who present in the UC San Diego Surgical Specialties clinic and have been cleared by the Bariatric and Metabolic Institute (BMI) team for bariatric surgery will be evaluated for participation in this trial. If the inclusion and exclusion criteria are met, the patients will be offered participation in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
To assess outcomes related to the transvaginal NOTES approach to laparoscopic sleeve gastrectomy (through data collection). | 1 year

SECONDARY OUTCOMES:
To assess pain associated with the transvaginal NOTES approach to laparoscopic sleeve gastrectomy (through data collection). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, M.D., FACS, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States